CLINICAL TRIAL: NCT03534531
Title: Prospective Observational Trial of Intra-Articular Cervical Zygapophyseal Joint Corticosteroid Injections in Patients With Increased Peri-Zygapophyseal Joint MRI Short Tau Inversion Recovery Signal
Brief Title: Cortisone Shots for Neck Pain
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Joshua Levin, Clinical Assistant Professor, Stanford University
Other Study IDs: IRB-45400
Record Dates: First submitted 2018-04-26; First posted 2018-05-23 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Neck Pain; Cervicalgia; Facet Joint Pain
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Intra-articular cervical zygapophyseal joint injection — Fluoroscopically-guided intra-articular cervical zygapophyseal steroid injection

SUMMARY:
The purpose of this study is to determine if cortisone shots in the neck are helpful in patients with certain MRI findings. Additionally, the investigators hope to learn if cervical facet joint steroid injections are beneficial in the subset of patients with MRI findings consistent with facet joint synovitis.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years old
* Patient who will be getting a neck cortisone shot for pain that has been there for at least 4 weeks
* A specific MRI finding (increased Short Tau Inversion Recovery signal) around 1 or more of the joints in the neck

Exclusion Criteria:

* Those receiving disability, worker's compensation, or are involved in litigation related to their pain.
* Those unable to read English and complete the assessment instruments.
* Those unable to attend follow up appointments
* The patient is incarcerated.
* Grade 2 or greater spondylolisthesis at the involved or adjacent segments.
* History of prior posterior cervical surgery. Anterior cervical surgery is not an exclusion criteria.
* Progressive motor deficit, and/or clinical signs of myelopathy.
* Prior neck cortisone shots within the past 6 months.
* Possible pregnancy or other reason that precludes the use of fluoroscopy.
* Allergy to contrast media or local anesthetics.
* BMI>35.
* Systemic inflammatory arthritis (e.g., rheumatoid arthritis, ankylosing spondylitis, lupus).
* Active infection or treatment of infection with antibiotics within the past 7 days.
* Chronic widespread pain or somatoform disorder (e.g. fibromyalgia).
* Addictive behavior, severe clinical depression, or psychotic features.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will be done on patients with neck pain who have a specific MRI finding. Patients who are at least 18 years old and have had neck pain for at least 4 weeks may be eligible.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2018-07-19 (Actual); Primary Completion 2023-11-26 (Actual); Study Completion 2023-11-26 (Actual)

PRIMARY OUTCOMES:
Change in Numeric Pain Rating Scale | Baseline, 2-4 weeks, and 3 months
  0 to 10 scale grading severity of pain

SECONDARY OUTCOMES:
Neck Disability Index | Baseline, 2-4 weeks, and 3 months
  Measure of neck pain related disability, scored between 0-50 with 0 being no disability and higher numbers being higher levels of disability
Work status | Baseline, 2-4 weeks, and 3 months
  Yes or No explaining if the patient is working
Medication use | Baseline, 2-4 weeks, and 3 months
  Yes or No explaining if the patient is taking pain medication
Use of other treatments | Baseline, 2-4 weeks, and 3 months
  Yes or No explaining if the patient is using other health care resources
Global Assessment of Change | 2-4 weeks and 3 months
  Question asking if the patient is improved, the same, or worse

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Stanford University, Palo Alto, California
  - Stanford University, Redwood City, California
  - Vanderbilt University, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No